CLINICAL TRIAL: NCT03550352
Title: Cannabinoids in People Living With HIV on Effective Antiretroviral Therapy: A Pilot Study to Assess Safety, Tolerability and Effect on Immune Activation
Brief Title: Cannabinoids in PLWHIV on Effective ART
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: expiration of study product; end of study product availability
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Tilray (Industry); CIHR Canadian HIV Trials Network (Network); Université du Québec a Montréal (Other); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Principal Investigator, Cecilia Costiniuk, MD, MSc, FRCPC, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTNPT 028; 2018-4336 (Registry Identifier: MUHC Research Ethics Board)
Record Dates: First submitted 2018-05-23; First posted 2018-06-08 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: HIV Infections
Keywords: HIV; Cannabinoids; HIV reservoir; Microbiome; CBD; THC; Inflammation; Immune activation
MeSH Terms: conditions — HIV Infections; Inflammation | interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1) THC and CBD combined (Experimental): TN-TC11M2 oral capsules (THC 2.5 mg / CBD 2.5 mg)
  Interventions: Drug: TN-TC11M2 oral capsules (THC 2.5 mg/CBD 2.5 mg)
- 2) CBD alone (Experimental): TN-C200M2 oral capsules (CBD 200 mg)
  Interventions: Drug: TN-C200M2 oral capsules (CBD 200 mg)

INTERVENTIONS:
Drug: TN-TC11M2 oral capsules (THC 2.5 mg/CBD 2.5 mg) — Participants will start by taking 1 capsule twice daily for 1 week (5 mg THC/5 mg CBD) and increase the number of capsules as tolerated to a maximum of 6 capsules taken throughout the day by weeks 5-12 (15 mg THC/15 mg CBD total per day).
  Arms: 1) THC and CBD combined
Drug: TN-C200M2 oral capsules (CBD 200 mg) — Participants will start by taking 1 capsule once daily for 1 week (200 mg CBD) and increase the number of capsules as tolerated to a maximum of 4 capsules taken throughout the day by weeks 5-12 (800 mg CBD total).
  Arms: 2) CBD alone

SUMMARY:
The purpose of this pilot study is to assess feasibility and to examine whether oral cannabinoids (capsules containing either Δ9-tetrahydrocannabinol (THC) and cannabidiol (CBD) combined or CBD alone) are safe and well-tolerated in people living with HIV. Other aims are to determine whether oral cannabinoids may reduce HIV-associated inflammation. An exploratory objective is to determine whether oral cannabinoids may influence HIV persistence as well as the gastrointestinal microbiome.

DETAILED DESCRIPTION:
Adults with well-controlled HIV (viral load suppressed for at least 3 years on effective antiretrovirals) will be randomized to receive Tilray oral capsules containing either THC and CBD (THC 2.5 mg / CBD 2.5 mg; TN-TC11M2) vs. CBD alone (CBD 200 mg; TN-C200M2). Participants will titrate up the number of capsules consumed based on their own individual tolerability, to a specified maximum daily dose, for a total treatment duration of 12 weeks.

Participants will be assessed regularly via history and physical exam as well as through safety blood work monitoring (hematology and chemistry profiles, liver enzymes, renal function, HIV viral loads, CD4 and CD8 counts). Effect on mood and quality of life will be determined by WHO-QOL-HIV-BREF, EQ-5D and Profile of Mood States questionnaires. Blood work for immune activation and inflammatory profiles, as well as HIV reservoir, will also be drawn at regular intervals.

This pilot study will provide information on feasibility (ie, time to recruitment of participants, whether participants continue the study for the full 12 week duration and complete the follow-up visits and questionnaires, whether treatment is safe and well-tolerated). It will also provide some preliminary data on the ability of TN-TC11M2 and TN-C200M2 oral capsules to reduce inflammation and possibly influence HIV persistence.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria within 4 weeks prior to the week 0 (Baseline 1) visit to be considered eligible for entry into the study:

  1. Documented HIV infection by Western Blot, EIA assays or viral load assays
  2. Male or female, Aged 18 or older
  3. Viral load <40 copies/ml for at least 3 years
  4. On ART for at least 3 years
  5. No cannabinoid use for at least 1 month prior to enrolment with negative baseline cannabinoid screen
  6. Able to communicate adequately in either French or English
  7. Able and willing to provide written informed consent prior to enrolment including access to relevant medical records

Exclusion Criteria:

1. Using cannabinoid-containing products outside of the study or within 4 weeks of study commencement
2. Pregnant, breastfeeding or planning to become pregnant during the course of the study. Female participants must undergo a pregnancy test and obtain a negative result in order to qualify for study participation.
3. Enrolled in a separate study involving administration of medication, vitamin, supplement or herbal product.
4. Active intravenous drug users
5. Active substance dependence
6. Prior history of hypersensitivity to cannabis or cannabis-containing products
7. Known or suspected allergy to sunflower lecithin oil
8. Active opportunistic infection or malignant condition
9. Unintentional weight loss of 10 % or more of body weight in the last 6 months
10. Unstable angina or acute cardiac event in the past year
11. Active psychiatric disorder or history of psychiatric depression (other than mild depression or anxiety); On antipsychotic medication
12. Known or suspected family history of schizophrenia or severe personality disorder
13. Serious cardiovascular disease such as ischemic heart disease, arrhythmias, poorly controlled hypertension, or severe heart failure
14. Anemia (Hemoglobin <100 g/L)
15. Active liver disease or unexplained persistent elevations of serum transaminases
16. Co-infection with Hepatitis B or C (positive HBsAg or positive anti-HBc antibodies with a detectable HBV DNA viral load or positive anti HCV antibodies with a detectable HCV RNA viral load)
17. Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) or alkaline phosphatase >2.5 x upper limit of normal (ULN)
18. Active AIDS event in the last month as determined by the treating physician
19. Renal dysfunction
20. Unstable psychological or psychiatric condition as determined by the treating physician
21. Holding employment which requires operation of heavy machinery or which requires undergoing drug screening (i.e., pilot or police officer)
22. Concurrent use within the past 8 week of anabolic hormones, prednisone, IL-2 or other agents known to alter immune function.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
WHO toxicity scale | week 0-12
  Proportions of participants in both groups without any signs of significant toxicity as determined by the WHO toxicity scale (i.e., number of participants with Grades 0-2 scores on the WHO toxicity scale) Proportion of participants in both groups without any signs of significant haematological, biochemical, hepatic, renal, cardiovascular, respiratory, gastrointestinal, neurological, musculoskeletal, dermatological or systemic toxicity (Grades 0-2) as determined by the World Health Organization Toxicity Grading Scale for Determining the Severity of Adverse events (Grades 0=no toxicity; Grade 1=mild, transient or mild discomfort vs. maximum score Grade 4=life-threatening, extreme limitation in activity, significant assistance required)
  Toxicity scores (Grade 0, 1, 2, 3, or 4) will be calculated and reported for each domain (hematology, biochemistry, hepatic enzymes, urinalysis, cardiovascular, respiratory, gastrointestinal, neurological, musculoskeletal, dermatological, systemic)

SECONDARY OUTCOMES:
Change in immune cell profile | week 0-12
  Change in CD4 count and their subsets including naïve, central memory and effector memory, Treg and Th17 cells from week 0 to week 12 Change in immune cell profile (frequencies of CD4 T cell counts and their subsets such as naïve, central memory and effector memory T cells; T regulatory cells; Th17 cells) from week 0 to week 12
Change in plasma inflammatory markers | week 0-12
  Change in plasma inflammatory markers from week 0 to week 12 Change in concentration of plasma inflammatory markers (interferon-α, interleukin-1β, interleukin-6, interleukin-10, interleukin-17, Transforming Growth Factor-β, interferon-gamma-induced protein-10, d-dimer, C-reactive protein, lipopolysaccharide and soluble CD14) from week 0 to week 12
Change in proportion activated CD4 and CD8 T cell lymphocytes | week 0-12
  Change in CD8+CD38+HLADR+ and CD4+CD38+HLADR+ percentages from week 0 to 12 weeks
  Change in proportion activated CD4 and CD8 T cell lymphocytes (CD38+HLADR+) from week 0 to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Costiniuk, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Chronic Viral Illnesses Service, McGill University Health Centre-Glen Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Costiniuk CT, Saneei Z, Routy JP, Margolese S, Mandarino E, Singer J, Lebouche B, Cox J, Szabo J, Brouillette MJ, Klein MB, Chomont N, Jenabian MA. Oral cannabinoids in people living with HIV on effective antiretroviral therapy: CTN PT028-study protocol for a pilot randomised trial to assess safety, tolerability and effect on immune activation. BMJ Open. 2019 Jan 17;9(1):e024793. doi: 10.1136/bmjopen-2018-024793. PMID 30659041